CLINICAL TRIAL: NCT06731010
Title: Non-invasive Neurophysiological Methods in Predicting and Evaluating Postoperative Pain in Patients Undergoing Major Thoracic Surgery
Brief Title: Application of Non-invasive Neurophysiological Methods in Predicting and Evaluating Postoperative Pain in Adult Patients Undergoing Major Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Chrysanthi Barba, Anaesthesiology Resident GH Evangelismos, National and Kapodistrian University of Athens
Other Study IDs: 298792022
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Pain, Acute; Postoperative Pain, Chronic; Postoperative Pain After Thoracic Surgery
Keywords: Postoperative pain; Pupillometry; EEG; Peak alpha frequency (PAF); Nociception Level Index (NOL)
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
The primary aim of this study is to explore the relationship between alpha electroencephalographic oscillations, particularly Peak Alpha Frequency (PAF), pupillometry, intraoperative Nociception Level (NOL) and postoperative pain following major thoracic surgeries.

Goals to investigate the use of preoperative EEG as a biomarker for the prediction of postoperative pain to investigate the use of pupillometry in postoperative pain prediction and evaluation to test intraoperative NOL as a predicting factor of postoperative pain

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older scheduled for open lung lobectomy due to early-stage lung cancer.

Exclusion Criteria:

* 1) Severe neurological disorders (e.g. dementia) that could interfere with EEG recordings or pain testing.

  2) Severe psychiatric conditions such as major depression, schizophrenia, or active drug abuse.

  3) Preoperative analgesic therapy, which may alter EEG signals (Boord et al. 2008).

  4) Diabetes mellitus 5) Chronic pain of any etiology 6) Acute pain from any cause

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Evangelismos General Hospital in Athens, Greece, for lung cancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | Pain intensity was recorded immediately postoperatively in the Post-Anesthesia Care Unit (PACU), as well as at 24, 48, and 72 hours after the surgery. Chronic postoperative pain was assessed both one month and three months after surgery.
  Pain intensity in patients was assessed postoperatively using the Numeric Rating Scale (NRS), specifically the Eleven-point NRS (NRS 0-10). Responses were categorized as follows: 0 : no pain, scores from 1 to 3 indicated mild pain, a score of 4-6 represented moderate pain, and scores of 7 or higher signified severe pain.Patients' postoperative late pain was assessed using NRS and the DN4 index. The DN4 (Douleur Neuropathique 4 questions) is a validated questionnaire used to diagnose neuropathic pain. It is utilized to evaluate postoperative pain and assess symptoms related to neuropathic pain, such as the spread of pain and alterations in sensory perception

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Evangelismos General Hospital, Athens, Attica
  - National and Kapodistrian University of Athens, Athens, Attica

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in publications: Only the individual-level data that directly support the published results or findings (e.g., data used in statistical analyses that led to conclusions). Anonymized data .
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Koschmieder KC, Funcke S, Shadloo M, Pinnschmidt HO, Greiwe G, Fischer M, Nitzschke R. Validation of three nociception indices to predict immediate postoperative pain before emergence from general anaesthesia: a prospective double-blind, observational study. Br J Anaesth. 2023 Apr;130(4):477-484. doi: 10.1016/j.bja.2022.11.024. Epub 2023 Jan 4. PMID 36609057
- [Background] Fang PP, Wu JQ, Tang LL, Gao S, Liu XS. The association between perioperative pupillary parameters and postoperative acute pain: A pilot cross-sectional study. Pain Pract. 2022 Mar;22(3):322-328. doi: 10.1111/papr.13084. Epub 2021 Oct 26. PMID 34662477
- [Background] Furman AJ, Prokhorenko M, Keaser ML, Zhang J, Chen S, Mazaheri A, Seminowicz DA. Sensorimotor Peak Alpha Frequency Is a Reliable Biomarker of Prolonged Pain Sensitivity. Cereb Cortex. 2020 Nov 3;30(12):6069-6082. doi: 10.1093/cercor/bhaa124. PMID 32591813
- [Background] Furman AJ, Meeker TJ, Rietschel JC, Yoo S, Muthulingam J, Prokhorenko M, Keaser ML, Goodman RN, Mazaheri A, Seminowicz DA. Cerebral peak alpha frequency predicts individual differences in pain sensitivity. Neuroimage. 2018 Feb 15;167:203-210. doi: 10.1016/j.neuroimage.2017.11.042. Epub 2017 Nov 21. PMID 29175204
- [Background] Millard SK, Furman AJ, Kerr A, Seminowicz DA, Gao F, Naidu BV, Mazaheri A. Predicting postoperative pain in lung cancer patients using preoperative peak alpha frequency. Br J Anaesth. 2022 Jun;128(6):e346-e348. doi: 10.1016/j.bja.2022.03.006. Epub 2022 Apr 4. No abstract available. PMID 35393099